CLINICAL TRIAL: NCT06288568
Title: Development and Evaluation of Nutritional Strategies to Reduce and Prevent Obesity in Shiftworkers
Brief Title: Night Shift Work and Biomarkers of Obesity Risk in Hospital and Industry Workers
Acronym: Shift2Health
Status: Recruiting | Type: Observational
Sponsor: University of Vienna (Other)
Collaborators: Medical University of Vienna (Other); FH Joanneum Gesellschaft mbH (Industry); Wageningen University and Research (Other); Wageningen University (Other); University of Bremen (Other); Verein zur Förderung des Technologietransfers an der Hochschule Bremerhaven e.V. (Unknown); UNIVERSYTET MEDYCZNY W LODZI (Unknown); Københavns Universitet (Other); Charite University, Berlin, Germany (Other); Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Karl-Heinz Wagner, Professor, University of Vienna
Other Study IDs: Shift2Health
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-02

CONDITIONS: Obesity; Shift-work Disorder; Circadian Rhythm Disorders
MeSH Terms: conditions — Obesity; Chronobiology Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Nightshift workers: Nightshift worker in the health care and industrial sector. Night shift is defined as a work schedule that involves working at least 3 hours between 00:00 and 5:00, at least 2 consecutive nights/month.
  Interventions: Other: No intervention
- Dayshift workers: Dayshift worker in the health care and industrial sector. No night shifts.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Shift work is a well-known risk factor for the development of overweight and obesity, which may lead to downstream effects such as increased risk of cardiometabolic diseases and cancer. However, the biological and behavioral mechanisms underlying the obesogenicity of night shift work are not well understood. Population-based mechanistic studies in real life shift workers are needed to address how night shift work impacts metabolic health.

The investigators aim to characterize the behavioural, environmental, and biological mechanisms and pathways for the association of night shift work and obesity across Europe.

The investigators will conduct a cross sectional study in 5 European countries (Austria, Denmark, Germany, Netherlands and Poland) and recruit 1000 rotating night shift workers and day workers (200/country) from the health sector and different industries. Night and day workers will be age-frequency (3 age groups), gender and (where possible) working tasks matched. Participants will complete online questionnaires and report their diet habits in a mobile app. Body composition, dietary behavior and sensory preferences will be tested. Biologic specimens (blood, urine, saliva, hair and feces) will be collected at the workplace on a day where participants are working on a day shift (or a day off). In a subsample (Austria and Netherlands) shift workers will provide biological samples (spot blood, urine and saliva) both on a day shift and on a night shift. Biomarkers including hormones, cellular immunity and inflammation, parameters linked to gut health and metabolism of fat and sugar, appetite, oxidative stress, metabolomics and microbiota will be measured. The investigators hypothesize that compared to day workers, night shift workers will experience disrupted levels of pre-obesity markers. Higher circadian disruption, sleep disruption and mistimed eating patterns workers will be associated with more disrupted biomarker profiles. Among rotating shift workers, night shift will be associated with acute disrupted melatonin production, metabolomic profiles and composition of oral microbiota compared to a day shift.

ELIGIBILITY:
Inclusion Criteria shift worker

* Health care sector or industrial shift worker
* Employed or self-employed
* 21 years or older
* ≥ 24 h/ week
* Shift work duration > 3 years and currently doing night shifts
* 4 or more rotating night shifts/month (night shift defined as a work schedule that involves working at least 3 hours between 00:00 and 5:00), at least 2 consecutive nights/month

Inclusion criteria controls

* Health care sector or industrial work
* Employed or self-employed
* 21 years or older
* ≥ 24 h/ week
* No night shift or rotating shift work in the last 5 years
* No history of night shift or rotating shift work for more than 5 years

Exclusion Criteria shift worker and controls:

* Pregnancy
* Lactation period
* BMI of 40 kg/m2 or above
* Present treatment of a disease e.g. cancer radio- or chemotherapy
* Chronic diseases if in an ongoing therapy but not after a remission (renal failure, active hepatitis, cirrhosis, myocardial infarction, chronic obstructive pulmonary disease and cancer)
* Immunodeficiency syndrome, any auto-immune or auto-inflammatory diseases (e.g. type-1 diabetes, multiple sclerosis, lupus, rheumatoid arthritis) and acute episodes of atopic diseases (atopic dermatitis, asthma, type 1 allergies such as hay fever)
* Bariatric surgery
* Antibiotics in the last month

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We are recruiting shift worker and day worker in the industrial and healthcare setting.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
high-sensitive C-Reactive Protein (hs-CRP) | Baseline
  Compare hs-CRP levels between night shift workers and day shift workers

SECONDARY OUTCOMES:
The investigators will consider levels of hormones in plasma | Baseline
  Compare melatonin levels between night shift workers and day shift workers
The investigators will consider levels of hormones in plasma | Baseline
  Compare cortisol levels between night shift workers and day shift workers
The investigators will consider levels of parameters linked to gut health in serum and in feces | Baseline
  Compare Short-chain fatty acids (SCFA) levels between night shift workers and day shift workers
The investigators will consider levels of parameters linked to gut health in serum and in feces | Baseline
  Compare Fatty acid-binding protein (FABP) levels between night shift workers and day shift workers
The investigators will consider levels of parameters linked to gut health in serum and in feces | Baseline
  Compare lipopolysaccharide(LPS)-binding protein levels between night shift workers and day shift workers
The investigators will consider levels of parameters linked to gut health in serum and in feces | Baseline
  Compare zonulin-1 levels between night shift workers and day shift workers
The investigators will consider parameters of cellular immunity and inflammation in plasma | Baseline
  Compare growth factors levels between night shift workers and day shift workers
The investigators will consider parameters of cellular immunity and inflammation in plasma | Baseline
  Compare cytokines levels between night shift workers and day shift workers
The investigators will consider parameters of cellular immunity and inflammation in plasma | Baseline
  Compare chemokines levels between night shift workers and day shift workers
The investigators will consider parameters of metabolism of fat and sugar in plasma | Baseline
  Compare total cholesterol levels between night shift workers and day shift workers
The investigators will consider parameters of metabolism of fat and sugar in plasma | Baseline
  Compare LDL-C levels between night shift workers and day shift workers
The investigators will consider parameters of metabolism of fat and sugar in plasma | Baseline
  Compare HDL-C levels between night shift workers and day shift workers
The investigators will consider parameters of metabolism of fat and sugar in plasma | Baseline
  Compare triglycerides levels between night shift workers and day shift workers
The investigators will consider parameters of metabolism of fat and sugar in plasma | Baseline
  Compare glucose levels between night shift workers and day shift workers
The investigators will consider levels of appetite markers in plasma | Baseline
  Compare leptin levels between night shift workers and day shift workers
The investigators will consider levels of appetite markers in plasma | Baseline
  Compare ghrelin levels between night shift workers and day shift workers
The investigators will consider levels of oxidative stress in whole blood, serum, plasma and urine | Baseline
  Compare DNA damage levels between night shift workers and day shift workers
The investigators will consider levels of oxidative stress in whole blood, serum, plasma and urine | Baseline
  Compare Malondialdehyde (MDA) levels between night shift workers and day shift workers
The investigators will consider levels of oxidative stress in whole blood, serum, plasma and urine | Baseline
  Compare 8-oxo-Guo/Gua levels between night shift workers and day shift workers
The investigators will consider levels of oxidative stress in whole blood, serum, plasma and urine | Baseline
  Compare protein carbonyls levels between night shift workers and day shift workers
The investigators will consider levels of oxidative stress in whole blood, serum, plasma and urine | Baseline
  Compare unconjugated bilirubin levels between night shift workers and day shift workers
The investigators will consider metabolomics analysis of plasma samples and dry blood spots (DBS) | Baseline
  Compare the levels of various metabolites between night shift workers and day shift workers
The investigators will consider microbiome analysis of feces samples and tongue swabs | Baseline
  Compare the levels of various microbiota composition between night shift workers and day shift workers

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria